CLINICAL TRIAL: NCT01909544
Title: Muscle Oxygenation and Metabolism in Response to a Localized Fatigue-inducing Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Muscle Metabolism and Oxygenation During Localized Fatigue-exercise in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Lung Association (Industry)
Responsible Party: Principal Investigator, Fernanda Ribeiro, PhD candidate, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MX-20665
Record Dates: First submitted 2013-07-16; First posted 2013-07-26 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Muscle fatigue; Energy metabolism; Muscle oxygenation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Experimental)
  Interventions: Other: Fatiguing exercise
- Room air (Sham Comparator)
  Interventions: Other: Fatiguing exercise

INTERVENTIONS:
Other: Fatiguing exercise — All participants (patients and healthy subjects) will perform the exercise both under normoxic (FiO2 = 0.21) and hyperoxic conditions (FiO2 = 100%)

SUMMARY:
The purpose of this study is to investigate whether a localized exercise, in which cardiorespiratory demand is reduced, will result in greater limb muscle fatigue in patients with COPD as a consequence of muscle oxygenation and muscle metabolism disturbances.

ELIGIBILITY:
Inclusion Criteria:

* COPD (FEV1/FVC < 0.70 and FEV1 < 0.80 predicted
* Healthy subjects: no evidence of airways obstruction (FEV1/FVC > 0.70 and FEV1 > 0.80 predicted)
* Smoking history > 15 pack-years

Exclusion Criteria:

* Chronic hypoxemia and/or hypercapnia (PaO2 < 60 mmHg or SpO2 < 88% at rest and/or PaCO2 > 45 mmHg)
* Recent exacerbation (< 3 months)
* Recent cancer (< 3 years)
* Diabetes
* Myopathy, neuromuscular or articular disease
* Unstable cardiac disease
* Absolute contraindications to exercise testing
* Regular physical activity or exercise training program in the last 2 months
* Physical activity score > 9 in the Voorips questionnaire
* Thigh skinfold thickness > 15 mm
* BMI > 30

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Muscle deoxygenation | 45 seconds post-exercise (knee-extension repetitions)
  Changes of deoxyhemoglobin/myoglobin concentrations measured by near-infrared spectroscopy of vastus lateralis muscle.
Muscle metabolism | 45 seconds post-exercise (knee extension repetitions)
  Changes in glycolytic and oxidative metabolism pathway markers, energy substrates (glycogen and glucose), end-products of glycolysis (pyruvate, and lactate), intermediate markers of glycolysis and high-energy phosphate compounds obtained from muscle biopsies

SECONDARY OUTCOMES:
Ventilatory response | Baseline, beginning and end of each serie of knee extensions (fatiguing exercise)
  Minute ventilation will be monitored during the fatigue-inducing exercise and it will be compared between subjects and conditions (FiO2 = 21% vs. FiO2 = 100%)
Quadriceps muscle fatigue | baseline, 15 min and 40 min after the fatigue-inducing exercise
  Quadriceps muscle fatigue will be determined by loss of quadriceps strength measured by magnetic stimulation after the fatigue-inducing exercise.
  Surface electromyography will also be measured to characterize muscle fatigue.
total muscle work | end of fatiguing exercise
  Total muscle work performed during fatigue-inducing exercise that will be composed by subsequent isokinetic knee-extensions repetitions at 40% of maximal peak torque

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada